CLINICAL TRIAL: NCT04733651
Title: A Randomized, Open-labelled and Controlled Clinical Trial to Investigate the Clinical Efficacy of Isoquercetin in the Treatment of Mild-to-moderate Hospitalised COVID-19 Patients
Brief Title: Study to Investigate the Clinical Efficacy of Isoquercetin in Patients With COVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nepal Health Research Council (Other Government)
Responsible Party: Principal Investigator, Dr. Pradip Gyanwali,MD, Director, Nepal Health Research Council
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-2021
Record Dates: First submitted 2021-01-31; First posted 2021-02-02 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — isoquercitrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (Active Comparator): In this arm subjects will receive the hospital COVID-19 standard care
  Interventions: Drug: Hospital standard of care for COVID-19
- Isoquercetin arm (Experimental): In this arm subjects will receive the hospital COVID-19 standard care + Isoquercetin
  Interventions: Drug: Hospital standard of care for COVID-19; Drug: Isoquercetin

INTERVENTIONS:
Drug: Hospital standard of care for COVID-19 — Standard care for COVID-19 as per the hospital guidelines
Drug: Isoquercetin — Daily 1000 mg Isoquercetin as 4 capsules
  Arms: Isoquercetin arm

SUMMARY:
The purpose of this study is to investigate the clinical efficacy of Isoquercetin in preventing disease progression and symptoms improvement in mild-to-moderate hospitalised COVID-19 patients.

DETAILED DESCRIPTION:
This is an open-labelled, randomized and multi-centre clinical trial in subjects with RT-PCR confirmed SARS-CoV-2 infection with mild-to-moderate symptoms, and who are currently admitted to the hospital for diagnosis of COVID-19. The study has two arms: hospital standard COVID-19 care (Control group) and hospital standard COVID-19 care + Isoquercetin (Isoquercetin group). The recruited subjects will be placed into either group by an electronic randomization process. Patients in the Isoquercetin group will receive a daily dose of 1000 mg Isoquercetin as 4 x 250 mg Isoquercetin capsules as add-on therapy in addition to the hospital standard COVID-19 care. The Isoquercetin treatment will continue for 28 days.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years and above.
2. Confirmed SARS-CoV-2 infection by PCR/RT-PCR. Patients with positive point of care tests can be randomised but have to be confirmed for SARS-CoV-2 by RT-PCR.
3. Presence of symptoms consistent with COVID-19 (e.g. shortness of breath, cough, sputum, muscle aches, headache, fatigue, sore throat, loss or change to sense of smell and/or taste, rhinorrhoea and anorexia).
4. WHO 10-point Clinical Progression Scale score of 4 to 5
5. Patient requires hospitalisation due to severity of COVID-19 or comorbidities if score 3 on the WHO 10-point Clinical Progression Scale.
6. Frailty score of ≤6.
7. Patient able to provide informed consent.
8. Females of child-bearing potential must be non-lactating, must have a negative pregnancy test at Screening, and must agree to continue using contraception throughout the study and for 4 weeks after study completion.

Exclusion Criteria:

1. Severe or critical COVID-19, e.g.:

   * Respiratory rate ≥ 30 breaths per minute OR
   * Heart rate ≥ 125 beats per minute OR
   * Respiratory failure, defined as clinical need for high-flow oxygen therapy, non- invasive positive pressure ventilation or endotracheal intubation and mechanical ventilation OR
   * Shock, defined as systolic blood pressure <90 mm Hg or diastolic blood pressure <60 mm Hg or requiring vasopressors OR
   * Multi-organ dysfunction/failure (WHO Clinical Progression Scale score ≥6)
2. Hospitalisation for reasons other than severity of COVID-19 or comorbidities (e.g. social reasons, local policies, isolation/quarantine).
3. Active bleeding or high risk for bleeding (e.g. known acute gastrointestinal ulcer).
4. History of significant haemorrhage (requiring hospitalisation or transfusion) outside of a surgical setting within the last 24 months.
5. Familial bleeding diathesis.
6. Glucose-6-phosphate dehydrogenase deficiency.
7. Severe hepatic and renal impairment as no safety and PK data of isoquercetin are available in these populations.
8. Current daily use of aspirin (> 81 mg daily), Clopidogrel (Plavix), cilostazol (Pletal), aspirin-dipyridamole (Aggrenox) (within 10 days) or considered to use regular use of higher doses of non-steroidal anti-inflammatory agents as determined by the treating physician (e.g. ibuprofen > 800 mg daily or equivalent).
9. Concomitant use of Cyclosporine, Warfarin (Coumarin), TPA, strong inducer of CYP3A4, or substrate of CYP3A4 with narrow therapeutic index.
10. History of allergic reactions attributed to compounds of similar chemical or biologic composition to isoquercetin.
11. Pregnancy.
12. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with isoquercetin, breastfeeding should be discontinued if the mother is treated with Isoquercetin. These potential risks may also apply to other agents used in this study.
13. Known hypersensitivity to Isoquercetin, Quercetin, or to any of the excipients used in the Isoquercetin capsules.
14. Patient with history of poor compliance, or current or past psychiatric disease that might interfere with the ability to comply with the study procedures or give informed consent according to the judgment of the investigator or institutionalized by court decision.
15. Patient with any condition that the physician judges could be detrimental to patient participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2021-02-20 (Estimated); Primary Completion 2021-05-20 (Estimated); Study Completion 2021-08-15 (Estimated)

PRIMARY OUTCOMES:
Disease progression, defined as WHO Clinical Progression Scale score of ≥ 6, at any time from day 1 to day 28 | From day 1 to day 28

SECONDARY OUTCOMES:
Disease recovery, defined as WHO Progression Scale score of ≤ 2, at day 28 | Day 1 through Day 28

OTHER OUTCOMES:
Change in the WHO Progression Scale score from baseline | Day 1 through Day 28
Changes in daily breathlessness, cough and sputum scale (BCSS) score (including disaggregated scores) | Day 1 through Day 28
Percentage of patients who progress to require mechanical ventilation | Day 1 through Day 28
Percentage of patients admitted to intensive care unit admission | Day 1 through Day 28
Time to recovery | Day 1 through Day 28
Time to hospital discharge | Day 1 through Day 28
Change in National Early Warning Score (NEWS 2) from baseline | Day 1 through Day 28
All-cause mortality | Day 1 through Day 28
QoL (EQ-5D-5L respiratory questionnaire) | Day 1 through Day 28

IPD SHARING:
Plan to Share IPD: No